CLINICAL TRIAL: NCT03887130
Title: Randomised Phase II Study of the Combination of Oral Vinorelbine With Capecitabine Versus Gemcitabine in Combination With Paclitaxel Versus Gemcitabine in Combination With Docetaxel as First Line Chemotherapy in Patients With Metastatic Breast Cancer
Brief Title: Study of Oral Vinorelbine Plus Capecitabine Versus Taxane-gemcitabine Combinations as 1st Line Chemotherapy in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM0259CA223B0
Record Dates: First submitted 2016-10-03; First posted 2019-03-22 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Capecitabine; Gemcitabine; Paclitaxel; Docetaxel

ARMS (3):
- Vinorelbine-Capecitabine (arm A) (Experimental): oral vinorelbine (OV) with capecitabine (CAP)
  Interventions: Drug: oral vinorelbine; Drug: Capecitabine
- Gemcitabine-Paclitaxel (arm B) (Active Comparator): gemcitabine (GEM) in combination with paclitaxel (PAC)
  Interventions: Drug: Gemcitabine 1250 mg/m²; Drug: Paclitaxel
- Gemcitabine-Docetaxel (arm C) (Active Comparator): gemcitabine (GEM) in combination with docetaxel (DOC)
  Interventions: Drug: Gemcitabine 1000 mg/m²; Drug: Docetaxel

INTERVENTIONS:
Drug: oral vinorelbine — Oral vinorelbine 60 mg/m² on day 1 & day 8, for cycle 1, and then 80 mg/m² on day 1 & day 8, every 3 weeks for subsequent cycles
  Arms: Vinorelbine-Capecitabine (arm A)
Drug: Capecitabine — Capecitabine 1000 mg/m² twice a day (2000 mg/m² daily) from day 1 to day 14
  Arms: Vinorelbine-Capecitabine (arm A)
Drug: Gemcitabine 1250 mg/m² — Gemcitabine 1250 mg/m² on day 1 & day 8
  Arms: Gemcitabine-Paclitaxel (arm B)
Drug: Gemcitabine 1000 mg/m² — Gemcitabine: 1000 mg/m² on day 1 & 8
  Arms: Gemcitabine-Docetaxel (arm C)
Drug: Paclitaxel — Paclitaxel 175 mg/m² on day 1
  Arms: Gemcitabine-Paclitaxel (arm B)
Drug: Docetaxel — Docetaxel 75 mg/m² on day 1
  Arms: Gemcitabine-Docetaxel (arm C)

SUMMARY:
The aim of this international open-label randomized phase II trial is to evaluate the efficacy and safety of an all-oral combination and two all-intravenous combinations as first-line therapy for HER2-negative mBC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the breast;
* Documented metastatic disease previously untreated by chemotherapy;
* HER2 negative (assessed by 0-1+ IHC or 2+ IHC with FISH-) on the primary tumor or on metastatic site;
* Karnofsky Performance Status 70%.

Exclusion Criteria:

* Local relapse alone after conservative treatment or contra-lateral tumor;
* Patients with symptoms suggesting CNS involvement or leptomeningeal metastases;
* Concomitant hormonal therapy for metastatic breast cancer;
* Prior chemotherapy in the metastatic setting;
* Patients previously treated with a vinca-alkaloid, capecitabine, gemcitabine or taxanes;
* Prior severe and unexpected reaction to fluoropyrimidine therapy (with or without documented DPD deficiency) or known hypersensitivity to 5-fluorouracil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2007-03-27 (Actual); Primary Completion 2013-04-18 (Actual); Study Completion 2013-04-18 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vinorelbine-Capecitabine (Arm A) | Gemcitabine-Paclitaxel (Arm B) | Gemcitabine-Docetaxel (Arm C)
Started | 51 | 50 | 51
Completed | 0 | 0 | 0
Not Completed | 51 | 50 | 51
Not completed — Progressive disease | 23 | 14 | 7
Not completed — Protocol Violation | 3 | 1 | 2
Not completed — Drug related toxicity | 7 | 7 | 13
Not completed — Non drug related toxicity | 3 | 0 | 0
Not completed — Death | 2 | 2 | 1
Not completed — Withdrawal by Subject | 7 | 6 | 11
Not completed — other reason | 6 | 20 | 17

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are described for the Intent-to-treat population that consisted of all treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Vinorelbine-Capecitabine (Arm A) | Gemcitabine-Paclitaxel (Arm B) | Gemcitabine-Docetaxel (Arm C) | Total
Number analyzed (Participants) | 49 | 50 | 50 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (9.7) | 56.0 (10.8) | 57.4 (9.7) | 56.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 50 | 50 | 149
  Male | 0 | 0 | 0 | 0
Body surface area [Mean (Standard Deviation); unit: mg/m²] | 1.8 (0.2) | 1.7 (0.2) | 1.8 (0.2) | 1.7 (0.2)
Delay between diagnosis and study entry [Mean (Standard Deviation); unit: years] | 5.5 (5.7) | 5.8 (6.3) | 5.8 (5.9) | 5.7 (5.9)
Primary tumour site [Count of Participants; unit: Participants]
  Bilateral | 3 | 0 | 0 | 3
  Left breast | 20 | 24 | 29 | 73
  Right breast | 26 | 26 | 21 | 73
Delay between first relapse/progression and study entry [Mean (Standard Deviation); unit: months] | 8.8 (19.1) | 11.1 (29.8) | 11.3 (23.9) | 10.4 (24.5)
Categorized number of organs involved at baseline [Count of Participants; unit: Participants]
  1 organ | 9 | 3 | 4 | 16
  2 organs | 14 | 25 | 17 | 56
  >= 3 organs | 26 | 22 | 29 | 77

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR)
Description: Disease control rate (DCR) defined as the sum of complete response, partial response and stable disease for at least 3 months according to RECIST criteria version 1.1.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI:
  Complete Response (CR)= Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
  Stable disease: no partial response or progression of the disease
Time Frame: From Baseline to disease progression or death, up to 6 years
Population: Disease control rate was measured in the Intent-to-treat ITT population that consisted of all treated patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vinorelbine-Capecitabine (Arm A) | Gemcitabine-Paclitaxel (Arm B) | Gemcitabine-Docetaxel (Arm C)
Number analyzed (Participants) | 49 | 50 | 50
percentage of participants | 73.5 [58.9 to 85.1] | 78.0 [64.1 to 88.5] | 80.0 [66.3 to 90.0]

ADVERSE EVENTS:
Time Frame: All adverse events were collected from the first dose of treatment through study completion up to 6 years
Arm/Group | Vinorelbine-Capecitabine (Arm A) | Gemcitabine-Paclitaxel (Arm B) | Gemcitabine-Docetaxel (Arm C)
All-Cause Mortality (participants affected / at risk) | 31/49 | 37/50 | 35/50
Serious Adverse Events (participants affected / at risk) | 13/49 | 16/50 | 12/50
Other Adverse Events (participants affected / at risk) | 49/49 | 50/50 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vinorelbine-Capecitabine (Arm A) (N=49) | Gemcitabine-Paclitaxel (Arm B) (N=50) | Gemcitabine-Docetaxel (Arm C) (N=50)
International normalised ratio (Investigations) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (2)
Malignant tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (4) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vinorelbine-Capecitabine (Arm A) (N=49) | Gemcitabine-Paclitaxel (Arm B) (N=50) | Gemcitabine-Docetaxel (Arm C) (N=50)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4)
Lacrimation increased (Eye disorders) | 3 (3) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 16 (16) | 6 (6) | 9 (9)
Abdominal pain upper (Gastrointestinal disorders) | 8 (8) | 3 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 7 (7) | 7 (7) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 29 (29) | 13 (13) | 19 (19)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 1 (1) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1)
Ileus (Gastrointestinal disorders) | 4 (4) | 4 (4) | 5 (5)
Nausea (Gastrointestinal disorders) | 29 (29) | 19 (19) | 22 (22)
Stomatitis (Gastrointestinal disorders) | 11 (11) | 4 (4) | 15 (15)
Vomiting (Gastrointestinal disorders) | 27 (27) | 12 (12) | 19 (19)
Chest pain (General disorders) | 3 (3) | 6 (6) | 4 (4)
Chills (General disorders) | 3 (3) | 2 (2) | 0 (0)
Fatigue (General disorders) | 38 (38) | 35 (35) | 42 (42)
Influenza like illness (General disorders) | 3 (3) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 6 (6) | 3 (3) | 13 (13)
Pain (General disorders) | 3 (3) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 6 (6) | 8 (8) | 13 (13)
Hypersensitivity (Immune system disorders) | 0 (0) | 5 (5) | 6 (6)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3) | 3 (3)
Neutropenic infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 6 (6) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 14 (14) | 7 (7) | 10 (10)
Weight increased (Investigations) | 3 (3) | 3 (3) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 19 (19) | 13 (13) | 17 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 15 (15) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6) | 2 (2)
Dizziness (Nervous system disorders) | 6 (6) | 2 (2) | 4 (4)
Dysgeusia (Nervous system disorders) | 1 (1) | 5 (5) | 11 (11)
Headache (Nervous system disorders) | 10 (10) | 8 (8) | 8 (8)
Paraesthesia (Nervous system disorders) | 5 (5) | 16 (16) | 4 (4)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (12) | 18 (18) | 8 (8)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (4) | 3 (3)
Depression (Psychiatric disorders) | 7 (7) | 4 (4) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (6) | 3 (3) | 3 (3)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 8 (8) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 13 (13) | 17 (17)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12) | 38 (38) | 40 (40)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 6 (6)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 24 (24) | 4 (4) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 11 (11) | 13 (13)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 1 (1) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 5 (5)
Hypotension (Vascular disorders) | 4 (4) | 2 (2) | 7 (7)
Lymphoedema (Vascular disorders) | 4 (4) | 2 (2) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No